CLINICAL TRIAL: NCT04420104
Title: Errector Spinae Plane Block for Postoperative Pain Management in Cardiac Surgery: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, Assoc. Prof. Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMU
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Erector Spinae Plane Block; Cardiac Surgery
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esp block group (Experimental)
  Interventions: Procedure: erector spinae plane block; Drug: iv analgesia
- control group (Active Comparator)
  Interventions: Drug: iv analgesia

INTERVENTIONS:
Procedure: erector spinae plane block — ESP Block: Bilateral ESP block and with ultrasound guidance will be applied A total 40 ml, 20 ml bupivacaine 0.5%, 20 ml saline.
  Arms: esp block group
Drug: iv analgesia — iv contromal

SUMMARY:
The purpose of this study is to assess efficacy of erector spinae plane block (ESP) for postoperative pain management in cardiac surgery patients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be randomised (single blind) as block group(patients is performed esp block) and control group. All patients will be evaluate during 48 hours for postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Must be ASA score I-III
* Must be 18-75 years old
* must undergo cardiac surgery

Exclusion Criteria:

* emergency surgery,
* bleeding diathesis,
* presence of contraindications to LA agents used in this study,
* use of chronic opioids,
* psychiatric disorders.
* prolonged extubation
* presence of infection at the injection site.
* cardiovascular conditions (EF<40, LMCA obstruction)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline in pain the 10 point Visual Analog Scale (VAS) at hours 3,6,9,12,24,36,48. | baseline and hours 3-6-12-24-36-48
  The VAS is validated instrument assessing average pain. Possible scores range from 0 (no pain) to 10 (worst possible pain) Change= (hours 3,6,9,12,24,48 score- baseline)
time to mobilize the patient | Any time for 7 days
  time to mobilize the patient is reported as when the patient is mobilized

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Sari, Assoc Prof, Principal Investigator — Adnan Menderes University Medical Faculty Hospital
Locations (1):
- Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991